CLINICAL TRIAL: NCT03491241
Title: Effect of Inflammatory Axis and Sirtuins' Expression in a Population of Overweight Pre-diabetics Patients From Metabolic Homeostasis Towards the Adipogonesis, and to Cardiac Redomelling.
Brief Title: Inflammatory Axis and Sirtuins' in Overweight Pre-diabetics Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Celestino Sardu, Principal investigator, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 22.3.2018
Record Dates: First submitted 2018-03-22; First posted 2018-04-09 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Pre-diabetes; Obesity
MeSH Terms: conditions — Glucose Intolerance; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- pre-diabetics obese patients (Experimental): These pre-diabetic obese patients will be treated by hypocaloric diet therapy. these patients were under metformine therapy at enrollment.
  Interventions: Dietary Supplement: hypocaloric diet therapy
- pre-diabetics patients (Placebo Comparator): These pre-diabetic patients will be treated by hypocaloric diet therapy alone.
  Interventions: Dietary Supplement: hypocaloric diet therapy
- obese patients (Active Comparator): These obese patients will be treated by hypocaloric diet therapy.
  Interventions: Dietary Supplement: hypocaloric diet therapy

INTERVENTIONS:
Dietary Supplement: hypocaloric diet therapy — all patients will receive an hypocaloric diet, with low carboidrates (<50%) overload.

SUMMARY:
In obese patients the superficial adipose tissue works as an endocrine active tissue to express different cytokines, and multiple molecular pathways implied in the cross talking with different part of the human body, such as the cardiovascular system. To date, adipocytes and adipose tissue-derived macrophages and adipose tissue synthesize, and secrete several cytokines, and sirtuins. In this setting, the excess of body fat is linked to heart contractile dysfunction. All these pathways are differently expressed in obese diabetic patients as compared to obese non diabetic patients. Intriguingly, in diabetic obese patients the hyper-expression of inflammatory cytokines is associated to a hypo-expression of sirtuins. Furthermore, microRNAs (miRs) as miR 195 and miR 27 could be implied in the regulation of this complex cellular and molecular axis.Therefore, this molecular pattern in diabetic obese patients may correlate to altered myocardial performance, and to the development of heart failure disease. In this study authors will evaluate at baseline by peripheral blood samples and by the abdominal fat tissue, and than at 12 months of follow-up by perupheral blood analysis, the expression of cytokines sirtuins and miR 195/27 comparing pre-diabetics obese patients vs. non pre-diabetics obese patients.

DETAILED DESCRIPTION:
In obese patients the visceral fat, and the superficial adipose tissue work as an endocrine active tissue to express different cytokines, and multiple molecular pathways implied in the cross talking with different part of the human body, such as the cardiovascular system. To date, adipocytes, and adipose tissue-derived macrophages and adipose tissue, synthesize and secrete several cytokines, like tumor necrosis factor (TNF)-5 and interleukin (IL)-6, and anti-apoptotic proteins, such as sirtuins. Sirtuins are NAD+-dependent deacetylase involved in the control of energy metabolism, adipocyte hypertrophy, and of different cardiac reparative, and rimodellative functions. Furthermore Sirtuins could cross talk with inflammatory/oxidative stress axis, and could be modulated by miR 195/27 expression. In this setting, the excess of body fat is linked to heart contractile dysfunction. It is intuitive to speculate that, all these pathways are differently expressed in obese diabetic patients as compared to obese non diabetic patients. Intriguingly, in diabetic obese patients the hyper-expression of inflammatory cytokines is associated to a hypo-expression of sirtuins, and over expression of miR 195 and miR 27. Therefore, this molecular pattern in diabetic obese patients may correlate to altered myocardial performance, and to the development of heart failure disease. Authors' study hypothesis is that, this complex altered bidirectional pattern between the inflammatory and apoptotic pathways axis may be due to a progressive increase in adipose tissue, produced by long-term alterations in energy balance. However, all these alterations may be measured in adipocytes as well as in adipose tissue derived macrophages, and by peripheral blood assay. Intriguingly, no data evaluated these pathways in pre-diabetics obese patients, and their possible correlation to cardiac function worsening, and to the development of heart failure disease. Actually, the pre-diabetic obese subjects represent a population of patients associated to higher risk to develop cardiovascular disease, myocardial dysfunction, and heart failure. In these patients a not clear indication exists about the right dietetic and/or drug treatment to control the hyperglycemia. However, there is discussion about the necessity or not to introduce hypoglycemic drug therapy added to a hypocaloric diet therapy to control the hyperglycemic overload. Therefore, the aim of the present study will be to evaluate at baseline the abdominal fat tissue expression of cytokines, sirtuins, miR 195 and miR 27 (by direct tissue biopsy) and by peripheral blood samples in pre-diabetics obese patients vs. non pre-diabetics obese patients. As second, during six and twelve months of follow up by peripheral blood samples analysis authors will evaluate the abdominal fat tissue expression of cytokines, miR 195 and miR 27 in pre-diabetics obese patients treated by hypocaloric diet-therapy as compared to pre-diabetics obese patients treated by hypocaloric diet-therapy plus metformine. At the end, authors will report their correlation to myocardial performance index (MPI) as an index of myocardial performance in pre-diabetics obese patients treated by hypocaloric diet-therapy as compared to pre-diabetics obese patients treated by hypocaloric diet-therapy plus metformine. Authors may speculate to observe a different cytokines, sirtuins, miR 195 and miR 27 expression at visceral fat and peripheral blood in pre-diabetics obese patients vs. non pre-diabetics obese patients. As second, authors may find that, hypoglycemic drug therapy may induce a down regulation of peripheral blood cytokines, a hyper expression of sirtuins, and a down regulation of miR 195 and miR 27 involved in the control of energy metabolism, and of adipocyte hypertrophy, and secondary implied in a better cardiac function at follow up.

ELIGIBILITY:
Inclusion Criteria:

* body mass index > 30;
* prediabetes;
* normal glycemic blood profile;
* both gender;
* age > 18 and < 65 years old.

Exclusion Criteria:

* body mass index < 30;
* diabetes;
* age < 18, and > 65 years old.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
left ventricle ejection fraction | 12 months
  authors will assess left ventricle ejection fraction by trans thoracic bidimensional echocardiographic measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- Raffaele Marfella, Naples, Italy

IPD SHARING:
Plan to Share IPD: Undecided